CLINICAL TRIAL: NCT00976105
Title: A Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of 10 Days of Repeat Dosing of GSK1521498 in Overweight or Obese But Otherwise Healthy Subjects.
Brief Title: Effects of Repeat Dosing of GSK1521498
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111849
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Obesity
Keywords: Pharmacokinetics; Pharmacodynamics; Safety and tolerability; Repeat dose; Personality traits; Fat mass; Healthy volunteers
MeSH Terms: conditions — Obesity | interventions — Zolpidem; N-((3,5-difluoro-3'-(1H-1,2,4-triazol-3-yl)-4-biphenylyl)methyl)-2,3-dihydro-1H-inden-2-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: Zolpidem or placebo (Active Comparator): This part is designed to examine the acute effects of up to 10mg of a known hypnotic sedative drug (Zolpidem) on cognitive and mood changes sensitve to sedation and tiredess.
  Interventions: Drug: Zolpidem or placebo - Hypnotic drug given for sleep disorders
- Part B: GSK1521498 or placebo (Experimental): At least 15 hours after Part A is completed subjects will enter Part B of the study.
  Interventions: Drug: GSK1521498 or placebo

INTERVENTIONS:
Drug: Zolpidem or placebo - Hypnotic drug given for sleep disorders — The information gathered from Part A will be used as a benchmark against which any effects of GSK1521498 can be assessed in Part B.
  Arms: Part A: Zolpidem or placebo
Drug: GSK1521498 or placebo — The first group will start at a low dose (10 mg GSK1521498 or placebo) for 10 days. The study team will then assess the data gathered from the first cohort and will select the dose that the next cohort will receive for 10 days. There will be up to 4 cohorts.
  Arms: Part B: GSK1521498 or placebo

SUMMARY:
The overall purpose of this study is to see whether the drug is safe and well tolerated when given to overweight or obese but otherwise healthy volunteers for 10 days. Up to 4 groups of people will be given the drug at variable strengths. The blood levels of the drug will be measured and the effects on mood and cognition (the mental processes involved in awareness, learning and judgement) will be assesed.

DETAILED DESCRIPTION:
This study is to test a new drug which may be used for treating eating behaviour and patterns that some overweight and obese patients find difficult to control. The drug works by inhibiting the effects of messenger molecules called opioids, e.g. endorphins. These opioids are naturally produced within the human body and control hunger, thirst, and the pleasurable feelings we relate to eating food. The drug attaches to opioid binding sites in the brain, known as mu-opioid receptors; this blocks the natural effect of opioids which may reduce the craving to eat fatty or sugary foods. Single doses of the drug have been given to humans and showed it was safe. Now the drug will be given every day for 10 days to check that the drug is safe and tolerated when given repeatedly. The study is in two parts:

Part A: people will receive a sleeping tablet to make them sleepy (or a dummy drug) and will complete some questionnaires and simple tests including computer exercises to test the effect of this tablet on mood and cognition. This information will be used to help judge what is happening in Part B.

Part B: requires staying in the unit for 10 days to receive a tablet every day and complete questionnaires and other tests to check for any mood and cognitive changes. Various other assessments will include effects on eating behaviour, pain measures and changes in body composition (content of fat, muscle and water).

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician
* Non smoking male or female between 18 and 60 years of age inclusive
* A female subject of child-bearing potential must use a contraception method listed in the protocol prior to the start of dosing until at least 14 days after receiving the last dose of study medication.
* Male subjects must agree to use one of the contraception methods listed in the protocol from the first dose of study medication until at least 84 days after receiving the last dose of study medication.
* BMI within the range 25 - 35 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF < 450 msec.
* Suitable for repeat cannulation.

Exclusion Criteria:

* Has clinically significant rhythm abnormalities identified during 24-hour screening Holter assessment.
* Systolic blood pressure greater than 150 mmHg and/or diastolic BP greater than 90 mmHg.
* Diabetes mellitus or physician-diagnosed dyslipidaemia requiring treatment
* Self-administered Beck Depression Inventory II scale total score greater than 13 or suicide question score greater than zero at screening.
* Positive pre-study drug/alcohol screen
* Positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Positive test for HIV antibody.
* Pregnant or lactating females
* Smoking history that includes regular use of tobacco or nicotine-containing products within 6 months prior to screening.
* A history of any thyroid dysfunction or an abnormal thyroid function test
* History of regular high level of alcohol consumption within 6 months of the study
* Participated in a clinical trial involving an investigational product within 90 days
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days prior to the first dose of study medication
* History of any gastrointestinal or hepatic conditions or procedures that could affect absorption of the investigational product.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that contraindicates participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol, including abstaining from consumption of caffeine-or xanthine containing products for 24 hours prior to dosing until the post-dose assessment, use of illicit drugs, refrain from alcohol for 24 hours prior to dosing until final post-dose assessment,, consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until after collection of the final pharmacokinetic blood sample.
* Any finding that would preclude safe use of Echo MRI scanning. These include: a history of panic attacks and/or claustrophobia, pacemaker, implanted hearing aid, metallic body piercing and/or other metal implants that cannot be removed, the opinion of the Investigator the subject exceeds size limitations for the instrument.
* Mentally or legally incapacitated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-09-22 (Actual); Primary Completion 2010-03-09 (Actual); Study Completion 2010-03-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: adverse events, blood pressure, heart rate, ECG, clinical chemistry, heamatology, urinalysis, change in reaction times, change in mood scales | During 10 days of repeat dosing
Obtain benchmarking data on the cognitive and mood changes induced by a single dose of up to 10mg zolpidem | Single occasion

SECONDARY OUTCOMES:
Assess accumulation, dose proportionality and pharmacokinetics of GSK1521498: AUC (0-24), Cmax, tmax, tlag (Dose 1 only), t1/2 (Dose 10 only), trough plasma concentrations on Day 5, 7, 8, 9 and 10 | On Day 1 and/or following 10 days of repeat dosing and trough samples on Day 5, 7, 8, 9 and 10
PK/PD relationships: cognitive and mood changes, pressure pain threshold and tolerance, heat pain threshold | During 10 days of reapeat dosing
Assess effects on body weight, fat mass, eating behaviour and personality traits: Bodyweight and BMI, Fat mass (ECHO-MRI), food ingested and energy intake, eating behaviour and persoality scales: Y-BOC-BE, BE, TFEQ and BIS | Screening, or Day -1 and Day 10

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111849 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111849?search=study&search_terms=111849#rs
- Available data/document: Individual Participant Data Set: 111849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111849 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register